CLINICAL TRIAL: NCT03547531
Title: Comparison of Modified Circular and Natural Tooth Brushing Methods in Effectiveness of Dental Plaque Removal in Children Aged 10-12 Years Old
Brief Title: Comparison of Modified Circular and Natural Tooth Brushing Methods in Effectiveness of Dental Plaque Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Istiyanti Hapsari, Comparison of Modified Circular and Natural Tooth Brushing Methods in Effectiveness of Dental Plaque Removal in Children Aged 10-12 Years Old, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5910820024
Record Dates: First submitted 2018-05-11; First posted 2018-06-06 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: the data were gathered from two groups of participants (control and intervention groups)
Who Masked: Outcomes Assessor
Masking Description: Examiner was blind to the allocation of the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Tooth Brushing Method (Active Comparator): Natural tooth brushing method is the method that is naturally used by the people with horizontal, rotary, or simple up and down motions and any position of the brush without any instruction of particular tooth brushing method.
  Interventions: Other: Natural Tooth Brushing Method
- Modified Circular Tooth Brushing Method (Experimental): Modified Circular tooth brushing method is a combination of small circular motion of brushing with the position of the brush slightly reach underneath the gingival that are applied for each jaw in all facial surfaces and posterior lingual of tooth arches.
  Interventions: Other: Modified Circular Tooth Brushing Method

INTERVENTIONS:
Other: Natural Tooth Brushing Method — Natural tooth brushing method is the method that is naturally used by the people with horizontal, rotary, or simple up and down motions and any position of the brush without any instruction of particular tooth brushing method.
  Arms: Natural Tooth Brushing Method
Other: Modified Circular Tooth Brushing Method — Modified Circular tooth brushing method is a combination of small circular motion of brushing with the position of the brush slightly reach underneath the gingival that are applied for each jaw in all facial surfaces and posterior lingual of tooth arches.
  Arms: Modified Circular Tooth Brushing Method

SUMMARY:
1. Plaque level in subjects using the Modified Circular method is different from that in subjects using natural tooth brushing method.
2. Gingivitis level in subjects using the Modified Circular method is different from that in subjects using natural tooth brushing method.
3. Level of plaque after using the Modified Circular method is different from that before using the method.
4. Level of gingivitis after using the Modified Circular method is different from that before using the method.

DETAILED DESCRIPTION:
Dental caries and gingivitis prevalences in schoolchildren in Indonesia is high. Dental diseases can potentially caused missed school, concentration disturbance, impaired speech, poor self-esteem, and systemic illness. Caries and gingivitis can be prevented by maintaining oral hygiene. Toothbrushing is one of oral hygiene method to remove and prevent dental plaque that can cause dental caries and gingivitis. The aim of the study was to compare the level of plaque and gingivitis of children aged 10-12 years old that use the Modified Circular and natural tooth brushing methods.

One hundred and twenty four students from two state elementary school in Yogyakarta, Indonesia participated in this study. The age of the participants were between 10 and 12 years old including males and females students. All of the participants were fifth graders from two elementary schools. To be eligible to participate in this study, each participants met the criteria including: students with age 10 to 12 years old and willing as well as permitted by the parents/guardian to join thorough the study. The exclusion criteria were being diagnosed having developmental disorder, using orthodontic appliances, and using antiseptic mouthwash for daily use.

The study began with the baseline data collection. Then it continued with the training for the participants about improving the oral hygiene. Children will be instructed to brush their teeth two times a day in the morning and before bedtime with the duration of 2 minutes. The project provided one toothpaste and one toothbrush for each children. In this stage, the intervention group was demonstrated and instructed to brush their teeth using Modified Circular method, while the control group was not given any instruction to brush their teeth using a specific tooth brushing method and asked to brush their teeth using the way they brushing every day. The period of intervention was started after training and lasted for one month. In intervention period, intervention group was observed once a week to ensure that they brushed their teeth correctly using Modified Circular method. Finally the evaluation was implemented after 1 month of intervention. The duration of the trial was one month, started in 2 August 2017 and finished on 6 September 2017, and the study was finished in time.

This study did not use any invasive treatment due to oral examination. No drugs or chemical materials were used except nontoxic disclosing agent that was used only 2-3 drops for staining the dental plaque. The colors of disclosing agent will gradually disapear and easily removed by brushing.

The benefit of this study was to help teachers, parents, and students to know the level of oral cleanliness and the effective method of toothbrushing in order to maintain oral hygiene and prevent dental caries and gingivitis.

The participants recruitment started after the research permission from government were accepted on 29 July 2017 until 31 July 2017. The schools selected then received the research permit from government and the research was started by giving the informed consent to the children and parents. The funding of this study is from Graduate School Prince of Songkla University Research Funding and Faculty of Dentistry Prince of Songkla University Research Funding.

The principle investigator of this study (as the main contact) is Istiyanti Hapsari (e-mail istiyantihapsari@gmail.com).

ELIGIBILITY:
Inclusion Criteria:

* Students with age 10 to 12 years old and willing as well as permitted by the parents/guardian to join thorough the study.

Exclusion Criteria:

* Being diagnosed having developmental disorder, using orthodontic appliances, and using antiseptic mouthwash for daily use.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Istiyanti Hapsari, Principal Investigator — Prince of Songkla University
Locations (1):
- Caturtunggal IV State Elementary School and Babarsari State Elementary School, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Data must be kept confidential to protect the privacy of participants. The shared data will be in the results in publication.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All of the participants were fifth graders from 2 elementary schools in Yogyakarta, Indonesia. These two schools have the similar characteristics in social-economy, number of students, and the type of school based on the data and recommendation from Education and Culture Office of Sleman District, Yogyakarta, Indonesia.
Pre-assignment Details: Each school had 62 fifth graders (total participants of both school was 124 fifth graders). No participants were excluded. Random group assignment was done by coin flipping to choose one school as control group and the other as intervention group.
Period: Overall Study
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method
Started | 62 | 62
Completed | 60 | 58
Not Completed | 2 | 4
Not completed — not coming in data collection : sick | 2 | 2
Not completed — having family occasion | 0 | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Number of teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method | Total
Number analyzed (Participants) | 62 | 62 | 124
Number analyzed (Number of teeth) | 1326 | 1328 | 2654
Age, Customized [Mean (Standard Deviation); unit: years]
  Age of participants | 10.9 (0.379) | 10.8 (0.342) | 10.8 (0.365)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Indonesia | 62 | 62 | 124

OUTCOME MEASURES:

1. Primary Outcome: Baseline Plaque Level
Description: Plaque level is examined using "Turesky Modification of Quigley-Hein Index". The scale is ranged from 0 to 5. 0 means no dental plaque existed on the tooth surface. 5 means all of the tooth surface is covered by dental plaque from the area that is closest to gingival to the occlusal area. The higher number of scores means worse. This index examines the buccal and lingual/palatal surfaces of the teeth (each teeth examined in 2 surfaces).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: plaque index
Units Other Than Participants: Number of teeth surfaces
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method
Number analyzed (Participants) | 62 | 62
Number analyzed (Number of teeth surfaces) | 2652 | 2656
plaque index | 2.25 (0.65) | 2.28 (1.68)
Statistical Analysis 1: Comparison: Natural Tooth Brushing Method vs Modified Circular Tooth Brushing Method; Null hypothesis: the mean of plaque index between groups are not different; Test type: Other; p > 0.05, t-test, 2 sided; independent t-test; the statistical analysis used in this study is independent t-test

2. Primary Outcome: Baseline Gingival Condition
Description: The examination of gingival condition was using the Gingival Index by Silness and Loe. A score between 0 and 3 was given based on the criteria:
  0= Normal gingiva.
  1. Mild inflammation - slight change in color, slight edema. No bleeding on probing.
  2. Moderate inflammation - redness, edema and glazing. Bleeding on probing.
  3. Severe inflammation - marked redness and edema. Ulceration. Tendency to spontaneous bleeding.
  This scale examine each teeth in 4 surfaces (mesial, distal, buccal, lingual/palatal).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: gingival index
Units Other Than Participants: Number of teeth surfaces
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method
Number analyzed (Participants) | 62 | 62
Number analyzed (Number of teeth surfaces) | 5304 | 5312
gingival index | 0.51 (0.28) | 0.49 (0.40)
Statistical Analysis 1: Comparison: Natural Tooth Brushing Method vs Modified Circular Tooth Brushing Method; null hypotesis: there is no difference of mean of gingival index between groups; Test type: Other — this data is analyzed using independent t-test; p > 0.05, t-test, 2 sided; this data is analyzed using independent t-test

3. Primary Outcome: Plaque Level at 1 Month
Description: as for outcome 1
Time Frame: one month after baseline data collection
Measure: Mean (Standard Deviation); unit: plaque index
Units Other Than Participants: Number of teeth surfaces
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method
Number analyzed (Participants) | 60 | 58
Number analyzed (Number of teeth surfaces) | 2564 | 2488
plaque index | 2.28 (1.19) | 1.68 (1.08)
Statistical Analysis 1: Comparison: Natural Tooth Brushing Method vs Modified Circular Tooth Brushing Method; null hypotesis: there is no difference of mean of plaque index between groups; Test type: Other — this data is analyzed using independent t-test; p < 0.05, t-test, 2 sided; this data is analyzed using independent t-test

4. Primary Outcome: Gingival Condition at 1 Month
Description: as for outcome 2
Time Frame: one month after baseline data collection
Measure: Mean (Standard Deviation); unit: gingival index
Units Other Than Participants: number of teeth surfaces
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method
Number analyzed (Participants) | 60 | 58
Number analyzed (number of teeth surfaces) | 5128 | 4976
gingival index | 0.49 (0.40) | 0.28 (0.33)
Statistical Analysis 1: Comparison: Natural Tooth Brushing Method vs Modified Circular Tooth Brushing Method; null hypotesis: there is no difference of mean of gingival index between groups; Test type: Other — this data is analyzed using independent t-test; p < 0.05, t-test, 2 sided; this data is analyzed using independent t-test

ADVERSE EVENTS:
Time Frame: Adverse events observation is done in final data collection which is collected in 1 month after the intervention to do Natural and Modified Circular tooth brushing methods given.
Description: no adverse events were found
Arm/Group | Natural Tooth Brushing Method | Modified Circular Tooth Brushing Method
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

LIMITATIONS AND CAVEATS:
Once a week observation in intervention group may cause the Hawthorne effect which was a consequence awareness of being studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03547531/Prot_SAP_ICF_000.pdf